CLINICAL TRIAL: NCT03445299
Title: Dementia and Sleep
Brief Title: Music for Dementia-related Sleep Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D&S2017
Record Dates: First submitted 2017-12-21; First posted 2018-02-26 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Dementia; Insomnia
MeSH Terms: conditions — Dementia; Sleep Initiation and Maintenance Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Within-subject design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music (Experimental): Daily music listening for 30 minutes at bedtime
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Music — Listening to music for 30 minutes at bedtime

SUMMARY:
The study aims to evaluate the effect of listening to music at bedtime on sleep in elderly persons with dementia and sleep problems.

DETAILED DESCRIPTION:
The study is a clinical trial to assess the effect of music listening as intervention for improving sleep in elderly persons with dementia and sleep problems. We use a within-subject design to evaluate the effect of the music intervention. Participants are persons above the age of 60 diagnosed with dementia and suffering from sleep problems. We will examine the effect of the intervention on sleep, mood and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Dementia
* Sleep problems

Exclusion Criteria:

* Use of hypnotic medications
* Substance abuse
* Severe hearing deficits
* Not out of bed during daytime

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Sleep | 14 days baseline and 14 days intervention
  Change in sleep pattern measured objectively with wrist actigraphy

SECONDARY OUTCOMES:
Sleep quality | After 14 days intervention period
  Change in sleep quality reported by primary caregiver (5 point Likert scale: 0=no change - 4=extreme change)
Depression | Measured at baseline and after 14 days intervention period
  Change in depressive symptoms as measured by the Geriatric Depression Scale (GDS). Scoring range 0-15. 0-4=no depression, 5-7=potential depression, >8=probable depression.
Cognition | Measured at baseline and after 14 days intervention period
  Change in cognitive functioning as measured by the Mini-Mental-State Examination (MMSE)
Mood | After 14 days intervention period
  Change in mood as reported by primary caregiver (5 point Likert scale: 0= no change - 4=extreme change)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Larsen, Study Chair — Technical University of Denmark
Locations (1):
- Center for Music in the Brain, Aarhus, Denmark